CLINICAL TRIAL: NCT02212964
Title: Differentiation of Pseudoprogression and True Progression Through High Field Susceptibility Weighted Imaging and R2*
Status: Completed | Type: Observational
Sponsor: Centre for Functional and Metabolic Mapping (Other)
Collaborators: London Regional Cancer Program, Canada (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: UWO105014
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Radiation Injury; Radiation Necrosis
Keywords: Radiation Injury; Radiation Necrosis; Ultra-high field MRI; Susceptibility Weighted Imaging; Post-treatment radiographic imaging change
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Using a multi-echo gradient echo sequence to calculate R2* and quantitative susceptibility maps and well as susceptibility-weighted imaging post processing the investigators hypothesize that the investigators would be able to distinguish between pseudoprogression and true progression with the use of an easily implementable sequence on clinical MRI scanners.

DETAILED DESCRIPTION:
Post-treatment radiographic imaging change (PTRIC) is seen in approximately 50% of patients who are treated for brain neoplasms using chemotherapy and radiotherapy. PTRIC can be attributed to true disease progression or a form of benign radiographic enhancement, known in literature as pseudoprogression. Of these patients, 50% of them have benign radiographic enhancement that is usually spontaneously resolved and required no intervention. The other 50% require immediate medical intervention, or more aggressive treatment for true progression. Currently standard medical practise is to administer a prophylactic treatment of chemotherapy to all patients with PTRIC with a follow up scan 3-6 months after initial PTRIC diagnosis, leading to up to 50% of patients receiving an unneeded dose of chemotherapy. The investigators hope to take advantage of the differentiation in tissue types and vascularization between true progression tumour and pseudoprogression to be able to identify patients who would not need to be administered a prophylactic dose of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must consent to participate.
2. The subject must be above the age of 18.
3. Patients must be classified as possible pseudoprogression or true progression
4. Patients scoring >= 70 on the karnofsky performance status.

Exclusion Criteria:

1. Any subject with contraindication to an MRI procedure as listed in the Magnetic Resonance Environment Screening Questionnaire.
2. Any subject who may be unable to tolerate the MRI environment due to physical size and/or known tendency to claustrophobia.
3. Any subject who does not expect to be available to attend the for the required study MRI scans
4. Patients scoring < 70 on the karnofsky performance status.
5. Attending radiation oncologist or neurologist determines patient is no longer able to consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had treatment for brain neoplasms treated with radiation and/or chemotherapy who presents with post-treatment imaging changes on the MRI following treatment.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 6 months
  R2* and susceptibility-weighted imaging venography to determine retrospectively if pseudoprogression can be distinguished from true progression

CONTACTS AND LOCATIONS:
Overall Officials: Ravi S Menon, PhD, Principal Investigator — Western University, Canada; Glenn Bauman, MD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada